CLINICAL TRIAL: NCT06514677
Title: A Comparison of Two Different Mechanical Interventions in Non-Surgical Peri-implantitis Treatment
Brief Title: Non-Surgical Treatment of Peri-Implantitis With Ultrasonic Carbon Tip
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Berceste Guler, Assoc Prof, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-13/01
Record Dates: First submitted 2024-07-15; First posted 2024-07-23 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Peri-Implantitis; Alveolar Bone Loss
MeSH Terms: conditions — Peri-Implantitis; Alveolar Bone Loss

STUDY DESIGN:
Intervention Model Description: Group I: Using Ultrasonic Carbon Tip for Non-surgical Peri-implantitis Treatment Group II: Using Titanium Curettes for for Non-surgical Peri-implantitis Treatment
Who Masked: Outcomes Assessor
Masking Description: For Outcomes Assessor Masking, Groups were not defined and anonymized and assessor will be blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasonic Carbon (Experimental): Using Ultrasonic Carbon Tip for Non-surgical Peri-implantitis Treatment
  Interventions: Procedure: Ultrasonic Carbon Tip
- Titanium (Active Comparator): Using Titanium Curettes for for Non-surgical Peri-implantitis Treatment
  Interventions: Procedure: Titanium Curette

INTERVENTIONS:
Procedure: Ultrasonic Carbon Tip — Using Ultrasonic Carbon Tip for Non-surgical Peri-implantitis Treatment
  Arms: Ultrasonic Carbon
Procedure: Titanium Curette — Using Titanium Curettes for for Non-surgical Peri-implantitis Treatment
  Arms: Titanium

SUMMARY:
As the frequency of dental implants increases, the incidence of complications and peri-implant diseases also increases. Early diagnosis and treatment of the disease is important to prevent consequences up to implant loss. Non-surgical treatment is the recommended treatment in the first stage due to its shorter duration and low morbidity rate. Non-surgical treatment of peri-implantitis provides clinical improvements such as reduced bleeding on probing (20-50%) and, in some cases, reduced pocket depth (≤ 1 mm). This study aims to clinically and radiographically compare two different mechanical treatments in patients with mild and moderate peri-implantitis.

DETAILED DESCRIPTION:
60 patients with at least one implant with mild to moderate peri-implantitis, defined as 2-4 mm radiographic reduced bone level, bleeding index (BI) ≥ 2, and probing pocket depth (PPD) ≥ 4 mm will be randomly allocated to test and control groups, receiving titanium curettes or ultrasonic Carbon tips debridement, respectively. Treatment was performed at baseline. Plaque index (PI), gingival index (GI), Periodontal pocket depth (PD), Bleeding on probing (BOP) gingival recession (GR) and Clinical attachment level (CAL) will be measured at four sites per implant and recorded by examiner at baseline, one, three, six and twelve months. Pus will be recorded as present/not present. The radiographic marginal bone level changes will be calculated at baseline, third months, sixth months and 12 months.

ELIGIBILITY:
Inclusion criteria:

1. Adult patients (≥18 years old)
2. Systemically healthy (ASA class 1 and ASA class 2)
3. Full-mouth plaque scores ≤20%
4. Implant had been in function for more than 6 months
5. Absence of plaque around the implant
6. Consent to complete all follow-up visits

Exclusion criteria:

1. Mobile implant
2. Overhanging restorations that prevent access to the implant for clinical measurements
3. Unresolvable technical complications that can cause peri-implantitis
4. Presence of active periodontal disease
5. Implants with a history of peri-implantitis treated using graft materials
6. Use of drugs that cause gingival hyperplasia
7. Systemic antibiotic use in the last 3 months
8. Acute and chronic medical conditions that prevent the patient from participating in the study
9. Presence of uncontrolled severe peri-implantitis from neighbouring implants
10. History of radiotherapy in the head and neck region
11. Receiving acute chemotherapy
12. Current corticosteroid therapy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Periodontal depth decrease | Baseline to 12th month
  Periodontal pocket depth (PD) decreasing baseline to 12th month

SECONDARY OUTCOMES:
marginal bone level changes | Baseline to 12th month
  Marginal bone level changes will be calculated at standardized periapical radiography

CONTACTS AND LOCATIONS:
Locations (1):
- Kütahya Health Sciences University Faculty of Dentistry, Department of Periodontology, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Linares A, Sanz-Sanchez I, Dopico J, Molina A, Blanco J, Montero E. Efficacy of adjunctive measures in the non-surgical treatment of peri-implantitis: A systematic review. J Clin Periodontol. 2023 Jun;50 Suppl 26:224-243. doi: 10.1111/jcpe.13821. Epub 2023 May 4. PMID 37143407
- [Background] Blasi A, Iorio-Siciliano V, Pacenza C, Pomingi F, Matarasso S, Rasperini G. Biofilm removal from implants supported restoration using different instruments: a 6-month comparative multicenter clinical study. Clin Oral Implants Res. 2016 Feb;27(2):e68-73. doi: 10.1111/clr.12530. Epub 2014 Dec 11. PMID 25496020
- [Background] Mensi M, Viviani L, Agosti R, Scotti E, Garzetti G, Calza S. Comparison between four different implant surface debridement methods: an in-vitro experimental study. Minerva Stomatol. 2020 Oct;69(5):286-294. doi: 10.23736/S0026-4970.20.04342-3. PMID 33174712
- [Background] Nart J, Pons R, Valles C, Esmatges A, Sanz-Martin I, Monje A. Non-surgical therapeutic outcomes of peri-implantitis: 12-month results. Clin Oral Investig. 2020 Feb;24(2):675-682. doi: 10.1007/s00784-019-02943-8. Epub 2019 May 23. PMID 31123873